CLINICAL TRIAL: NCT03662425
Title: Effects of Oxytocin on Negative Symptoms and Social Cognition in Schizophrenia and Its Behavioral Mechanisms
Brief Title: Effects of Oxytocin on Negative Symptoms and Social Cognition in Schizophrenia and Its Possible Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KLMH2018K02
Record Dates: First submitted 2018-06-27; First posted 2018-09-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia
Keywords: schizophrenia; negative symptoms; oxytocin
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- schizophrenia with oxytocin (Experimental): Participants self-administered the oxytocin twice daily via intranasal route: before breakfast and before dinner. Each dose consists of six 0.1 ml insufflations (alternating between the left and right nostril) of oxytocin spray containing approximately 24 international units of oxytocin.
  Interventions: Drug: Oxytocin
- schizophrenia with Placebo (Placebo Comparator): Participants self-administered the placebo twice daily via intranasal route: before breakfast and before dinner. Each dose consists of six 0.1 ml insufflations (alternating between the left and right nostril) of oxytocin spray containing approximately 24 international units of placebo.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Oxytocin — It's a two-week treatment trial.Subjects self-administer intranasal study drug twice daily; before breakfast and before dinner. Each dose consists of six 0.1 ml insufflations (alternating between the left and right nostril) of OT spray containing approximately 24 international units of OT
  Arms: schizophrenia with oxytocin
Drug: Saline — It's a two-week treatment trial. Subjects self-administer intranasal study drug twice daily; before breakfast and before dinner. Each dose consists of six 0.1 ml insufflations (alternating between the left and right nostril) of saline spray containing approximately 24 international units of saline
  Arms: schizophrenia with Placebo

SUMMARY:
The purpose of this study was to investigate the effects of oxytocin on negative symptoms and social cognitive task performance in schizophrenia. The investigators conducted a randomized, placebo-controlled trial testing the effects of twice daily intranasal oxytocin treatment for 14 days on psychotic symptoms and social cognition in patients with schizophrenia. The investigators hypothesize that PANSS scores will decline significantly and several social cognition measures will improved significantly or nearly significantly in oxytocin but not placebo recipients.

DETAILED DESCRIPTION:
Social impairment is a primary cause of disability in schizophrenia, responds poorly to current antipsychotic medications and is related to deficits in social cognitive abilities, which include Theory of Mind, emotion recognition and attributional style. Oxytocin (OT) has many pro-social effects in animals and antipsychotic-like efficacy in preclinical tests. In this study, the investigators conducted a randomized, placebo-controlled trial testing the effects of twice daily intranasal oxytocin treatment for 14 days on psychotic symptoms and social cognition in patients with schizophrenia. The investigators will recruit patients with schizophrenia, screening of subjects included a review of psychiatric and medical history, physical examination, baseline social cognition measures were obtained followed by psychiatric ratings. Daily intranasal treatments were initiated after baseline assessments. Social cognition measures and psychiatric ratings were repeated beginning 50 min after the morning dose of study medication on treatment day 14. psychiatric ratings include The Positive and Negative Syndrome Scale (PANSS) and The Clinical Assessment Interview for Negative Symptoms (CAINS). The social cognition instruments are some social scales such as Toronto Alexithymia Scale, the Interpersonal Reactivity Index(IRI), and some computer tests such as reinforcement learning task and facial emotion identification test.

ELIGIBILITY:
Inclusion criteria were:

1. aged between 18 and 55 years;
2. DSM-IV diagnosis of schizophrenia, acute schizophreniform disorder, or schizoaffective disorder.

Exclusion criteria were:

1. presence of other psychiatric diagnoses (e.g., depression);
2. active misuse of substance or alcohol;
3. intellectual disability (IQ < 70);
4. a history of neurological disorder.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-07-21 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | baseline
  The Positive and Negative Syndrome Scale (PANSS) is a 30-items, 7-point rating scale, the 7 rating points represent increasing levels of psychopathology, 7 were chosen to constitute Positive Scale, 7 items for Negative Scale and the remaining 16 items for a General Psychopathology Scale. The scale scores range from 30 to 210, with higher scores indicating more severe psychotic symptoms.
The Positive and Negative Syndrome Scale (PANSS) | the two-week endpoint
  The Positive and Negative Syndrome Scale (PANSS) is a 30-items, 7-point rating scale, the 7 rating points represent increasing levels of psychopathology, 7 were chosen to constitute Positive Scale, 7 items for Negative Scale and the remaining 16 items for a General Psychopathology Scale. The scale scores range from 30 to 210, with higher scores indicating more severe psychotic symptoms.
The Clinical Assessment Interview for Negative Symptoms (CAINS) | baseline
  The Clinical Assessment Interview for Negative Symptoms (CAINS) is used to assess negative symptoms, the CAINS is a 13-item interview-based assessment comprising a nine-item "motivation and pleasure" factor (items included recreation, social and vocational expected pleasure and motivation), and a four-item "expression" factor (items included vocal prosody, gestures, facial, and speech). All items were scored on a five-point scale from 0 (no impairment) to 4 (severe deficit).The scale scores range from 0 to 52, with higher scores indicating more severe negative symptoms.
The Clinical Assessment Interview for Negative Symptoms (CAINS) | the two-week endpoint
  The Clinical Assessment Interview for Negative Symptoms (CAINS) is used to assess negative symptoms, the CAINS is a 13-item interview-based assessment comprising a nine-item "motivation and pleasure" factor (items included recreation, social and vocational expected pleasure and motivation), and a four-item "expression" factor (items included vocal prosody, gestures, facial, and speech). All items were scored on a five-point scale from 0 (no impairment) to 4 (severe deficit).The scale scores range from 0 to 52, with higher scores indicating more severe negative symptoms.

SECONDARY OUTCOMES:
Reinforcement Learning Task | baseline
  The Gain versus Loss-Avoidance (GLA) task is a probabilistic reinforcement learning paradigm involving stimulus pairs in which choices resulted in reward or in loss avoidance.
Reinforcement Learning Task | the two-week endpoint
  The Gain versus Loss-Avoidance (GLA) task is a probabilistic reinforcement learning paradigm involving stimulus pairs in which choices resulted in reward or in loss avoidance.
The Temporal Experience of Pleasure Scale (TEPS) | baseline
  The Chinese version of the TEPS contains 20 items, using a 6-point Likert scale (from 1 = very false for me to 6 = very true for me), and measures anticipatory pleasure and consummatory pleasure, with higher scores indicating better pleasure experience.
The Temporal Experience of Pleasure Scale (TEPS) | the two-week endpoint
  The Chinese version of the TEPS contains 20 items, using a 6-point Likert scale (from 1 = very false for me to 6 = very true for me), and measures anticipatory pleasure and consummatory pleasure, with higher scores indicating better pleasure experience.
Interpersonal Reactivity Index (IRI) | baseline
  The Interpersonal Reactivity Index (IRI) (Davis, 1983) measures participants' empathic tendencies, it is a 28-item self-report scale measuring empathy and consists of four subscales: perspective taking, fantasy, personal distress, and empathic concern. While the first two subscales index, cognitive empathy, the last two subscales index affective empathy, each item is rated on a 5-point Likert scale ranging from 0 (does not describe me well) to 4 (describes me very well), and higher scores on the IRI-PT and the IRI-EC reflect greater cognitive and emotional empathy, respectively. In the Chinese version of the IRI, 6 items were deleted and 22 items remained (Chan, 1986) and it has been reported to have good reliability and validity in both normal and schizophrenic populations.
Interpersonal Reactivity Index (IRI) | the two-week endpoint
  The Interpersonal Reactivity Index (IRI) (Davis, 1983) measures participants' empathic tendencies, it is a 28-item self-report scale measuring empathy and consists of four subscales: perspective taking, fantasy, personal distress, and empathic concern. While the first two subscales index, cognitive empathy, the last two subscales index affective empathy, each item is rated on a 5-point Likert scale ranging from 0 (does not describe me well) to 4 (describes me very well), and higher scores on the IRI-PT and the IRI-EC reflect greater cognitive and emotional empathy, respectively. In the Chinese version of the IRI, 6 items were deleted and 22 items remained (Chan, 1986) and it has been reported to have good reliability and validity in both normal and schizophrenic populations.
Toronto Alexithymia Scale (TAS) | baseline
  The Toronto Alexithymia Scale (TAS-20) is used to assess the severity of alexithymia, it is a 20-item self-report instrument rated on a 5-point Liker-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 20 to 100, with higher scores indicating higher level of alexithymia. The TAS-20 consist of 3 factors: difficulty identifying feelings (DIF); difficulty describing feelings (DDF); externally oriented cognitive style of thinking (EOT). The Chinese version has been shown with having the same factor structure of the original version and has been associated with good internal consistency [15], which was adopted in this study.
Toronto Alexithymia Scale (TAS) | the two-week endpoint
  The Toronto Alexithymia Scale (TAS-20) is used to assess the severity of alexithymia, it is a 20-item self-report instrument rated on a 5-point Liker-type scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 20 to 100, with higher scores indicating higher level of alexithymia. The TAS-20 consist of 3 factors: difficulty identifying feelings (DIF); difficulty describing feelings (DDF); externally oriented cognitive style of thinking (EOT). The Chinese version has been shown with having the same factor structure of the original version and has been associated with good internal consistency [15], which was adopted in this study.
emotion recognition task | baseline
  The facial emotion identification test is used to assess facial emotion identification abilities, in which participants viewed 91 digital pictures of faces selected from the Japanese Female Facial Expression (JAFFE) Database (1998) and were asked to judge which emotion that particular face displayed on the screen was expressing (happy, sad, angry, afraid, surprise, disgusted or neutral).
emotion recognition task | the two-week endpoint
  The facial emotion identification test is used to assess facial emotion identification abilities, in which participants viewed 91 digital pictures of faces selected from the Japanese Female Facial Expression (JAFFE) Database (1998) and were asked to judge which emotion that particular face displayed on the screen was expressing (happy, sad, angry, afraid, surprise, disgusted or neutral).

CONTACTS AND LOCATIONS:
Overall Officials: Zhenghui Yi, Ph.D, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China